CLINICAL TRIAL: NCT00231972
Title: Enhancing HIV Prevention Among HIV Infected Men
Brief Title: Enhancing HIV Prevention by Using Behavioral Intervention Among HIV-Infected Men
Acronym: Enhance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Dr. Kenneth Mayer, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH068746 (NIH); DAHBR 9A-ASPG (Other: National Institute of Mental Health (NIMH-DAHBR)); R01MH068746 (NIH)
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: HIV; MSM
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project Enhance (Experimental): Participants will receive the risk reduction program, Project Enhance
  Interventions: Behavioral: Project Enhance
- Active Comparison Condition (Active Comparator): Participants will receive standard prevention case management
  Interventions: Behavioral: Standard prevention case management (PCM)

INTERVENTIONS:
Behavioral: Project Enhance — The behavioral intervention will be administered by a trained medical social worker on an individual basis. It will include an education component, as well as motivational and behavioral skills enhancement. Treatment will occur for only the first 3 months, after which follow-up sessions will be held every 3 months for the remainder of the year.
  Other Names: Project Enhance Behavioral Intervention
  Arms: Project Enhance
Behavioral: Standard prevention case management (PCM) — Participants will receive standard PCM for HIV prevention.
  Other Names: Project Enhance Prevention Case Management
  Arms: Active Comparison Condition

SUMMARY:
This study will evaluate the effectiveness of a behavioral intervention program versus standard prevention case management in promoting safer sex practices in HIV-infected men.

DETAILED DESCRIPTION:
In recent years, the spread of HIV and other STDs has increased, especially among men who have sex with men. This increase signifies continued sexual risk taking within this population. In order to curb the increase of HIV infections, prevention programs are needed. A standard prevention case management program has been developed; however, new programs that further improve outcomes are needed. This study will evaluate the effectiveness of a behavioral intervention program versus standard prevention case management (PCM) in promoting safer sex practices in HIV-infected men.

Participants in this 1-year open-label study will be randomly assigned to receive either PCM alone or a behavioral intervention called Project Enhance, in addition to PCM. The behavioral intervention will be administered by a trained medical social worker on an individual basis. It will include an education component, as well as motivational and behavioral skills enhancement. PCM will entail standard case management, as well as referrals to specific services that each individual may need. Treatment will occur for only the first 3 months, after which follow-up sessions will be held every 3 months for the remainder of the year.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Receives primary health care at Fenway Community Health
* Identifies as a man who has sex with men
* Has engaged in unprotected anal or vaginal intercourse within 3 months of study enrollment

Exclusion Criteria:

* All episodes of unprotected anal intercourse occurred with only a single primary partner who is also HIV infected
* Plans to relocate over the upcoming year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2003-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Reduction in rates of unprotected anal intercourse from baseline to 12-month follow-up | Measured at Months 3, 6, 9, and 12

SECONDARY OUTCOMES:
Incidence of sexually transmitted diseases | Measured at Months 3, 6, 9, and 12
Higher risk-reduction self-efficacy | Measured at Months 3, 6, 9, and 12
Increased behavioral intentions to engage in safer behaviors | Measured at Months 3, 6, 9, and 12
Increased risk-reduction strategies (other than condom use) | Measured at Months 3, 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mayer, MD, Principal Investigator — Fenway Community Health and Brown University; Steven Safren, PhD, Principal Investigator — Fenway Community Health and Harvard Medical School; Conall O'Cleirigh, PhD, Study Director — Fenway Community Health and Massachusetts General Hospital
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States